CLINICAL TRIAL: NCT06710158
Title: Phase Ⅰ Study to Evaluate the Safety/Tolerability, Pharmacokinetics, and Efficacy of SC-102 in Subjects With Advanced or Metastatic Solid Tumors That Express EphA2
Brief Title: Study of SC-102 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tianjin ConjuStar Biologics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SC-102-101
Record Dates: First submitted 2024-11-21; First posted 2024-11-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Cancers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SC-102 for once weekly (Experimental): Participants will receive SC-102 as a single agent once weekly on a 4-week cycle at the selected dose.
  Interventions: Drug: SC-102
- SC-102 for once biweekly (Experimental): Participants will receive SC-102 as a single agent once biweekly on a 4-week cycle at the selected dose.
  Interventions: Drug: SC-102

INTERVENTIONS:
Drug: SC-102 — SC-102 is a peptide drug conjugate (PDC) consisting an EphA2-targeting peptide, a tubulin inhibitor, and a protease-hydrolyzable linker.

SUMMARY:
This study will evaluate the safety, PK profile, and anti-cancer efficacy of SC-102 in subjects with advanced solid tumors

DETAILED DESCRIPTION:
SC-102 is a peptide drug conjugate (PDC) consisting of an EphA2-targeting peptide, a tubulin inhibitor, and a protease-hydrolysable linker.

This phase I multi-center, open-label first-in-human trial, including a dose escalation study and a dose expansion study, will evaluate SC-102 administrated once weekly or biweekly as a single agent in patients with advanced solid tumors. The dose escalation study is primarily designed to assess the safety and tolerability of SC-102 and to determine the recommended dose(s) for the dose expansion study. The dose expansion study is designed with the primary objective of evaluating the clinical activity of SC-102.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily agree to participate in the study and sign the Informed Consent Form (ICF).
2. Aged 18 to 75 years at the time of signature of the ICF, without gender limitation.
3. Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0 or 1.
4. Life expectancy of ≥ 3 months as assessed by the investigator.
5. Women and men of childbearing potential must be advised and agree to practice effective methods of contraception during the study.
6. Must be willing and able to comply with the protocol and study procedures.
7. Acceptable renal, hepatic, hematologic, and coagulation functions.
8. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
9. Metastatic recurrent histologically confirmed malignant solid tumors and exhausted all appropriate treatment options per local guidelines.
10. Confirmation of EphA2 expression by the central laboratory prior to enrollment is not required for participants enrolled in the dose escalation study, but required for participants enrolled in the dose expansion study.

Exclusion Criteria:

1. History of other malignancy(ies) within 3 years before signing the ICF, except for cured basal cell carcinoma or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, papillary carcinoma of the thyroid gland, carcinoma in situ of the duct in situ, or other malignant tumors that have survived without disease for more than 5 years.
2. Any anticancer treatment, including experimental treatments, within 4 weeks before the first dose of the study drug.
3. Radiotherapy to >30% of the bone marrow or extensive radiotherapy within 4 weeks, or local radiotherapy (e.g., radiation therapy to the thoracic spine and ribs) within 7 days, prior to the first dose of the study drug.
4. Uncontrolled central nervous system metastases.
5. Preexisting treatment-related toxicity Grade ≥ 2 (except Grade 2 alopecia and hypothyroidism stable with hormone replacement therapy).
6. Preexisting Grade ≥ 2 (as per CTCAE v5.0) sensory or motor neuropathy.
7. Major surgery within 4 weeks prior to the first dose of the study drug.
8. History of interstitial lung disease (ILD), preexisting ILD, or the suspected ILD that cannot be ruled out by imaging examination at screening.
9. Preexisting serious dermatological diseases, or having experienced serious skin toxicities during the prior anti-cancer treatment (e.g., Stevens-Johnson syndrome, toxic Epidermal Necrolysis, etc.).
10. Active infection requiring systemic therapy within 14 days prior to the first dose of the study drug.
11. History of thromboembolic events and bleeding disorders ≤ 3 months (e.g., deep vein thrombosis (DVT) or pulmonary embolism (PE)) prior to the first dose of the study drug.
12. Positive results of virus serology tests.
13. History of serious cardiovascular and cerebrovascular diseases.
14. Has received treatment within 2 weeks prior to the first dose of the study drug, or requires ongoing treatment with a medication that is a strong inhibitor or inducer of the cytochrome P450 3A4 (CYP3A4) enzymes.
15. Known sensitivity to any of the ingredients of the investigational product.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Number of participants receiving SC-102 treatment with treatment-emergent adverse events (escalation study) | From Cycle 1 Day 1 (each cycle is 28 days) until 30 days post last dose
  Safety reported as incidence of treatment-emergent adverse events
Maximum tolerated dose (MTD) by the number of participants with dose limiting toxicities from SC-102 treatment (escalation study) | At the end of Cycle 1 (each cycle is 28 days)
  Maximum Tolerated Dose (MTD)
Objective response rate by RECIST 1.1 in participants with solid tumors receiving SC-102 treatment (expansion study) | From Cycle 1 Day 1 (each cycle is 28 days) until the date of first documented progression, death from any cause, start treatment of new anti-cancer agent(s), loss of follow-up, or withdrawal of consent, which ever came first, assessed up to 2 years
  Defined as the percentage of subjects who experience a best response of either complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of SC-102 and monomethyl auristatin E (MMAE) | From Cycle 1 Day 1 through the end of treatment from any cause, assessed up to 2 years
  Plasma concentrations of SC-102 and MMAE from all participants receiving SC-102 treatment
Minimum plasma concentration (Cmin) of SC-102 and monomethyl auristatin E (MMAE) | From Cycle 1 Day 1 through the end of treatment from any cause, assessed up to 2 years
  Plasma concentrations of SC-102 and MMAE from all participants receiving SC-102 treatment
Area under the plasma concentration-time curve (AUC) of SC-102 and monomethyl auristatin E (MMAE) | From Cycle 1 Day 1 through the end of treatment from any cause, assessed up to 2 years
  Plasma concentrations of SC-102 and MMAE from all participants receiving SC-102 treatment
Elimination half-life (t1/2) of SC-102 and monomethyl auristatin E (MMAE) | From Cycle 1 Day 1 through the end of treatment from any cause, assessed up to 2 years
  Plasma concentrations of SC-102 and MMAE from all participants receiving SC-102 treatment
Number of participants positive for anti-drug antibodies (ADA) | From Cycle 1 Day 1 through the end of treatment from any cause, assessed up to 2 years
  Number of participants positive for anti-drug antibodies (ADA) from all participants receiving SC-102 treatment
Duration of Response (DoR) | From Cycle 1 Day 1 (each cycle is 28 days) until the date of first documented progression or death from any cause, which ever came first, assessed up to 2 years
  Defined as the time from first assessment of partial response (PR) or complete response (CR) until disease progression.
Disease Control Rate (DCR) | From Cycle 1 Day 1 (each cycle is 28 days) until the date of first documented progression, death from any cause, start treatment of new anti-cancer agent(s), loss of follow-up, or withdrawal of consent, which ever came first, assessed up to 2 years
  Defined as the percentage of subjects who experience a best response of either complete response (CR), partial response (PR), or stable disease (SD).

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No